CLINICAL TRIAL: NCT00738660
Title: Efficacy of Telmisartan and the Combination of Telmisartan and Ramipril in type1 Diabetes Patients With Nephropathy
Acronym: START1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sanjay K Bhadada, Post graduaate institute of medical education and research
Organization: PIMERIndia (Unknown)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: START1DM
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Diabetic Nephropathy
Keywords: type1 DM; microalbuminuria; nephropathy; albumin excretion rate; dual blockade; ACEI; ARB
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Diseases | interventions — Telmisartan; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): single experimental arm cross over of patients, addition of Ramipril onto Telmisartan.
  Interventions: Drug: Telmisartan, Ramipril

INTERVENTIONS:
Drug: Telmisartan, Ramipril — 80 mg of telmisartan administered for 8weeks,followed by addition of ramipril 10 mg for further 8weeks
  Other Names: cardace; cardiopri; tazloc

SUMMARY:
Hypothesis:

The angiotensin receptor blocker telmisartan is effective at reduction of albumin excretion rate(AER) in patients with type1 diabetes and micro or macroalbuminuria. Dual blockade with the addition of ramipril an angiotensin receptor blocker gives added efficacy for reduction of AER. ARB telmisartan gives a 24 hr BP lowering effect.

Summary:

This is an open label cross over study involving 30 patients who were initially treated with Telmisartan 80 mg for eight weeks followed by addition of Ramipril 10 mg for a further eight weeks. Albuminuria reduction and BP reduction with both clinic and ambulatory BP records were studied at the end of each phase.

DETAILED DESCRIPTION:
To evaluate the antialbuminuric efficacy of an angiotensin receptor blocker (ARB) telmisartan and the combination of telmisartan and ramipril in patients with type1 DM and either micro or macroalbuminuria.To evaluate the same drugs for their antihypertensive efficacy and their influence on dipping patterns using ambulatory BP monitoring.

Methods:

Open label cross over study involving 30 patients who were initially treated with telmisartan 80 mg for eight weeks followed by addition of ramipril 10 mg for a further eight weeks. Albuminuria reduction and BP reduction with both clinic and ambulatory BP records were studied at the end of each phase Overnight urine samples of nine hours duration were collected . The volume of urine was verified by measurement in a jar with accuracy of 50ml by the study investigator on every occasion. . Albuminuria was estimated by immuno-turbidimetry Hemocue albumin system Angelholm AD, Sweden (inter assay CV 4.3% ). The albumin excretion rate(AER) at baseline evaluation was determined as the mean AER of the positive urine samples. During subsequent evaluations at the end of 8weeks and at the end of 16 weeks the mean albumin excretion rate from two successive overnight urine samples was taken as the mean .Ambulatory BP (ABP) measurement :ABP was measured using Spacelabs device 90207 Spacelabs inc. use of which is described before(14) .A uniform protocol of inflation once in every 30 min was used. Cuff was applied to the nondominant arm. Recordings were started in all patients between seven and ten AM.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus by ADA criteria
* Clinical history of DKA
* HbA1C < 7.5,urine AER >/= 20 mcg/min on two overnight urine samples

Exclusion Criteria:

* Pregnancy
* Unwillingness to use contraception during time of study
* Creatinine >3 mg/dl
* Suspected/proven non diabetic nephropathy
* Active urinary sediment

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduction in albumin excretion rate | 8 weeks

SECONDARY OUTCOMES:
24 hr ambulatory BP reduction,nocturnal BP reduction, proportion of dippers | 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: sanjay k bhadada, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India